CLINICAL TRIAL: NCT02166463
Title: A Randomized Phase 3 Study of Brentuximab Vedotin (SGN-35) for Newly Diagnosed High-Risk Classical Hodgkin Lymphoma (cHL) in Children and Young Adults
Brief Title: Brentuximab Vedotin and Combination Chemotherapy in Treating Children and Young Adults With Stage IIB, Stage IIIB, IVA, or IVB Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCI-2014-01223; NCI-2014-01223 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s15-00950; AHOD1331 (Other: Children's Oncology Group); AHOD1331 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Results first posted 2023-05-31 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-06

CONDITIONS: Ann Arbor Stage IIB Hodgkin Lymphoma; Ann Arbor Stage IIIB Hodgkin Lymphoma; Ann Arbor Stage IVA Hodgkin Lymphoma; Ann Arbor Stage IVB Hodgkin Lymphoma; Childhood Hodgkin Lymphoma; Classic Hodgkin Lymphoma
MeSH Terms: interventions — Bleomycin; Brentuximab Vedotin; Cyclophosphamide; Doxorubicin; Etoposide; Methylprednisolone; exifone; Medrol Veriderm; Prednisone; deltacortene; prednylidene; Vincristine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (ABVE-PC) (Active Comparator): Patients receive doxorubicin hydrochloride IV over on days 1-2, bleomycin sulfate IV or SC on days 1 and 8, vincristine sulfate IV on days 1 and 8, etoposide IV on days 1-3, prednisone orally PO BID or methylprednisolone IV on days 1-7, and cyclophosphamide IV on days 1 and 2. Treatment repeats every 21 days for 5 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bleomycin Sulfate; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Methylprednisolone; Other: Pharmacological Study; Drug: Prednisone; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Vincristine Sulfate
- ARM II (Bv-AVEPC) (Experimental): Patients receive brentuximab vedotin IV on day 1. Patients also receive doxorubicin hydrochloride, etoposide, prednisone or methylprednisolone, and cyclophosphamide as in Arm I and vincristine sulfate IV on day 8. Treatment repeats every 21 days for 5 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Methylprednisolone; Other: Pharmacological Study; Drug: Prednisone; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Vincristine Sulfate

INTERVENTIONS:
Biological: Bleomycin Sulfate — Given IV or SC
  Other Names: Blanoxan; BleMomycine; Blenoxane; Bleo-cell; Bleo-S; Bleocin; Bleolem; Bleomycin Sulfas; Bleomycin Sulphate; Bleomycini Sulfas; Blexane; Oil Bleo
  Arms: Arm I (ABVE-PC)
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN 35; SGN-35; SGN35
  Arms: ARM II (Bv-AVEPC)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Methylprednisolone — Given IV
  Other Names: Adlone; Caberdelta M; DepMedalone; Depo Moderin; Depo-Nisolone; Duralone; Emmetipi; Esametone; Firmacort; Medlone 21; Medrate; Medrol; Medrol Veriderm; Medrone; Mega-Star; Meprolone; Methylprednisolonum; Metilbetasone Solubile; Metrocort; Metypresol; Metysolon; Predni-M-Tablinen; Prednilen; Radilem; Sieropresol; Solpredone; Summicort; Urbason; Veriderm Medrol; Wyacort
Other: Pharmacological Study — Correlative studies
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase III trial studies brentuximab vedotin and combination chemotherapy to see how well they work compared to combination chemotherapy alone in treating children and young adults with stage IIB with bulk, stage IIIB, IVA, or IVB Hodgkin lymphoma. Combinations of biological substances in brentuximab vedotin may be able to carry cancer-killing substances directly to Hodgkin lymphoma cells. Chemotherapy drugs, such as doxorubicin hydrochloride, bleomycin sulfate, vincristine sulfate, etoposide, prednisone, and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known if combination chemotherapy is more effective with or without brentuximab vedotin in treating children with high-risk Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the event free survival (EFS) of a novel regimen incorporating brentuximab vedotin (Bv; Adcetris) in the chemotherapy backbone of doxorubicin hydrochloride (doxorubicin) (Adriamycin), vincristine sulfate (vincristine), etoposide, prednisone and cyclophosphamide (Bv-AVEPC) in newly diagnosed high-risk classical Hodgkin lymphoma (cHL) compared to those treated with Adriamycin, bleomycin sulfate, vincristine sulfate, etoposide, prednisone, and cyclophosphamide (ABVE-PC).

SECONDARY OBJECTIVES:

I. To determine whether children/young adults with high-risk cHL treated with Bv-AVEPC have a higher rate of early response (determined by fludeoxyglucose F 18 [FDG]-positron emission tomography [PET]) and a reduction in protocol directed radiation therapy (RT) compared to those treated with ABVE-PC.

II. To compare the rate of neuropathy (>= grade 3) among patients treated on the Bv-AVEPC (experimental arm) to patients treated on the ABVE-PC (standard arm).

EXPLORATORY OBJECTIVES:

I. To validate and compare the Childhood Hodgkin International Prognostic Score (CHIPS) to conventional Ann Arbor stage (stages II B with bulk, III B, IV A or B) in predicting outcome in high-risk childhood cHL.

II. To determine the incidence of preferentially expressed antigen in melanoma (PRAME) and testis-specific antigens in Epstein-Barr virus (EBV)- cHL tumors and the incidence of EBV antigens (Epstein-Barr nuclear antigen 1 [EBNA1], Epstein-Barr virus latent membrane protein 1 [LMP1], large multifunctional peptidase 2 [LMP2]) in EBV+ cHL tumors, with the goal of developing strategies to integrate cellular therapy into treatment for newly diagnosed high-risk cHL. (Biology) III. To incorporate qualitative visual FDG-PET into response-directed treatment algorithms and explore quantitative FDG-PET and computed tomography (CT) definitions of tumor burden and response for incorporation into next generation pediatric cHL risk-stratification schemes, exploring the extension of these algorithms to young adults. (Imaging) IV. To evaluate the reduction in normal tissue irradiation associated with the current treatment approach compared to the volume of historic involved field radiation therapy (IFRT) fields. (Radiation Therapy) V. To evaluate EFS and patterns of relapse following protocol-specified RT utilization and treatment volumes. (Radiation Therapy) VI. To characterize the extent of chemotherapy induced peripheral neuropathy (CIPN), as reported by patients and parent proxies, through serial administration of the Functional Assessment of Cancer Therapy-Gynecologic Oncology Group-Neurotoxicity (FACT-GOG-NTX). (Patient Reported Outcomes [PRO] of Peripheral Neuropathy and Health-Related Quality of Life) VII. To describe the Health-Related Quality of Life (HRQL) consequences of peripheral neuropathy over time by correlating total neuropathy scale scores with the individual items with the Child Health Ratings Inventories (CHRIs)-Global scale (e.g., physical health, pain, emotional functioning). (PRO of Peripheral Neuropathy and Health-Related Quality of Life) VIII. To perform a cross validation of the FACT-GOG-NTX with the Total Neuropathy Score-Pediatric Vincristine (TNS-PV) to determine the performance of both measures with the use of brentuximab vedotin in a limited institutional approach in children and adolescents with cHL. (PRO of Peripheral Neuropathy and Health-Related Quality of Life) IX. To assess the resource use and cost implications of Bv in combination with chemotherapy and radiotherapy (RT) for newly diagnosed high-risk cHL in children and young adults. (Economic) X. To estimate the risk of relapse among rapidly responding lesions (RRL) subjects that have at least one lesion that is Deauville 3 at PET 2. (Follow-up of Deauville score 3 lesions on FDG-PET imaging [confirmed by central imaging review]) XI. To characterize the pharmacokinetics of brentuximab vedotin in children < 13 years of age.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I (ABVE-PC): Patients receive doxorubicin hydrochloride intravenously (IV) over on days 1-2, bleomycin sulfate IV or subcutaneously (SC) on days 1 and 8, vincristine sulfate IV on days 1 and 8, etoposide IV on days 1-3, prednisone orally (PO) twice daily (BID) or methylprednisolone IV on days 1-7, and cyclophosphamide IV on days 1 and 2.

ARM II (Bv-AVEPC): Patients receive brentuximab vedotin IV on day 1. Patients also receive doxorubicin hydrochloride, etoposide, prednisone or methylprednisolone, and cyclophosphamide as in Arm I and vincristine sulfate IV on day 8.

In both arms, treatment repeats every 21 days for 5 cycles in the absence of disease progression or unacceptable toxicity. Granulocyte simulating factor (GCSF) or equivalent is given on both arms.

After completion of study treatment, patients are followed up at 3, 6, 9, 12, 18, 24, 30, 36, and 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed, pathologically confirmed cHL meeting one of the following Ann Arbor stages are eligible:

  * Stage IIB with bulk
  * Stage IIIB
  * Stage IVA
  * Stage IVB

    * If study eligibility by staging is uncertain, consultation with Imaging and Radiation Oncology Core (IROC) Rhode Island (RI) may be obtained prior to study enrollment
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows (performed within 14 days prior to enrollment):

  * 2 to < 6 years: male 0.8 mg/dL, female 0.8 mg/dL
  * 6 to < 10 years: male 1 mg/dL, female 1 mg/dL
  * 10 to < 13 years: male 1.2 mg/dL, female 1.2 mg/dL
  * 13 to < 16 years: male 1.5 mg/dL, female 1.4 mg/dL
  * >= 16 years: male 1.7 mg/dL, female 1.4 mg/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (performed within 14 days prior to enrollment)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate transaminase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine transaminase [ALT]) < 2.5 x upper limit of normal (ULN) for age (performed within 14 days prior to enrollment)
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by radionuclide angiogram
* Forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) > 60% by pulmonary function test (PFT), unless due to large mediastinal mass from Hodgkin lymphoma (HL)
* For children who are unable to cooperate for PFTs, the criteria are: no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry reading of > 92% on room air
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with nodular lymphocyte-predominant HL
* Patients with an immunodeficiency that existed prior to diagnosis, such as primary immunodeficiency syndromes, organ transplant recipients and children on current systemic immunosuppressive agents are not eligible
* Patients who are pregnant; (since fetal toxicities and teratogenic effects have been noted for several of the study drugs, a negative pregnancy test is required for female patients of childbearing potential)
* Lactating females who plan to breastfeed
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation and for 30 days after the last dose of chemotherapy
* Patients known to be positive for human immunodeficiency virus (HIV) are not eligible
* Patients who have received any previous chemotherapy or radiation therapy are not eligible
* Patients who received systemic corticosteroids within 28 days of enrollment on this protocol, except as specified, are not eligible

Ages: 2 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2026-10-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Castellino, Principal Investigator — Children's Oncology Group
Locations (199):
- United States (182):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (14):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Puerto Rico (3):
  - HIMA San Pablo Oncologic Hospital, Caguas
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Toner K, Renfro LA, Dave H, Pezzella G, Pei Q, Giulino-Roth L, Horton T, Keller FG, Kelly KM, Castellino SM, Bollard CM. Tumor-specific immune responses and biomarkers in pediatric patients with high-risk Hodgkin lymphoma. Blood Adv. 2026 Jan 13;10(1):183-191. doi: 10.1182/bloodadvances.2025016797. PMID 40990939
- [Derived] Williams AM, Rodday AM, Renfro LA, Wu Y, Henderson TO, Keller FG, Punnett A, Hodgson D, Kelly KM, Castellino SM, Parsons SK. Group-based trajectories of health-related quality of life among pediatric patients with high-risk Hodgkin lymphoma. J Natl Cancer Inst. 2025 Oct 1;117(10):2112-2119. doi: 10.1093/jnci/djaf197. PMID 40700618
- [Derived] Tie X, Shin M, Lee C, Perlman SB, Huemann Z, Weisman AJ, Castellino SM, Kelly KM, McCarten KM, Alazraki AL, Hu J, Cho SY, Bradshaw TJ. Automatic Quantification of Serial PET/CT Images for Pediatric Hodgkin Lymphoma Using a Longitudinally Aware Segmentation Network. Radiol Artif Intell. 2025 May;7(3):e240229. doi: 10.1148/ryai.240229. PMID 39969278
- [Derived] Pabari R, McCarten K, Flerlage J, Lai H, Mauz-Korholz C, Dieckmann K, Palese M, Kaste S, Castellino SM, Kelly KM, Stoevesandt D, Kurch L. Hodgkin lymphoma involving the extra-axial CNS: an AHOD1331, PHL-C1, and PHL-C2 report from the COG and EuroNet-PHL. Blood Adv. 2024 Sep 24;8(18):4856-4865. doi: 10.1182/bloodadvances.2023012346. PMID 39058968
- [Derived] Williams AM, Rodday AM, Pei Q, Henderson TO, Keller FG, Punnett A, Kelly KM, Castellino SM, Parsons SK. Longitudinal Health-Related Quality of Life Among Patients With High-Risk Pediatric Hodgkin Lymphoma Treated on the Children's Oncology Group AHOD 1331 Study. J Clin Oncol. 2024 Oct;42(28):3330-3338. doi: 10.1200/JCO.24.00038. Epub 2024 Jul 26. PMID 39058966
- [Derived] Parsons SK, Rodday AM, Pei Q, Keller FG, Wu Y, Henderson TO, Cella D, Kelly KM, Castellino SM. Performance of the FACT-GOG-Ntx to assess chemotherapy-induced peripheral neuropathy (CIPN) in pediatric high risk Hodgkin lymphoma: report from the Children's Oncology Group AHOD 1331 study. J Patient Rep Outcomes. 2023 Nov 10;7(1):113. doi: 10.1186/s41687-023-00653-0. PMID 37947987
- [Derived] Castellino SM, Giulino-Roth L, Harker-Murray P, Kahn JM, Forlenza C, Cho S, Hoppe B, Parsons SK, Kelly KM; COG Hodgkin Lymphoma Committee. Children's Oncology Group's 2023 blueprint for research: Hodgkin lymphoma. Pediatr Blood Cancer. 2023 Sep;70 Suppl 6(Suppl 6):e30580. doi: 10.1002/pbc.30580. Epub 2023 Jul 28. PMID 37505794
- [Derived] Hoppe BS, McCarten KM, Pei Q, Kessel S, Alazraki A, Mhlanga JC, Lai HA, Eutsler E, Hodgson DC, Roberts KB, Charpentier AM, Keller FG, Voss SD, Wu Y, Cho SY, Kelly KM, Castellino SM. Importance of Central Imaging Review in a Pediatric Hodgkin Lymphoma Trial Using Positron Emission Tomography Response Adapted Radiation Therapy. Int J Radiat Oncol Biol Phys. 2023 Aug 1;116(5):1025-1030. doi: 10.1016/j.ijrobp.2023.02.020. Epub 2023 Mar 2. PMID 36868525
- [Derived] Castellino SM, Pei Q, Parsons SK, Hodgson D, McCarten K, Horton T, Cho S, Wu Y, Punnett A, Dave H, Henderson TO, Hoppe BS, Charpentier AM, Keller FG, Kelly KM. Brentuximab Vedotin with Chemotherapy in Pediatric High-Risk Hodgkin's Lymphoma. N Engl J Med. 2022 Nov 3;387(18):1649-1660. doi: 10.1056/NEJMoa2206660. PMID 36322844
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (ABVE-PC) | ARM II (Bv-AVEPC)
Started | 300 | 300
Completed | 262 | 273
Not Completed | 38 | 27
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 10 | 10
Not completed — Ineligible | 11 | 2
Not completed — Progressive Disease | 9 | 6
Not completed — Repeat eligibility studies are outside the parameters required for eligibility | 2 | 2
Not completed — Patient enrollment onto another COG study with tumor therapeutic intent | 1 | 0
Not completed — Refusal of further protocol therapy | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (ABVE-PC) | ARM II (Bv-AVEPC) | Total
Number analyzed (Participants) | 300 | 300 | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 285 | 290 | 575
  Between 18 and 65 years | 15 | 10 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (3) | 14.8 (3.1) | 15 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 139 | 281
  Male | 158 | 161 | 319
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 63 | 120
  Not Hispanic or Latino | 228 | 220 | 448
  Unknown or Not Reported | 15 | 17 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 9 | 7 | 16
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 33 | 34 | 67
  White | 221 | 224 | 445
  More than one race | 0 | 5 | 5
  Unknown or Not Reported | 34 | 27 | 61
Region of Enrollment [Number; unit: participants]
  United States | 281 | 277 | 558
  Canada | 19 | 23 | 42

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival (EFS), Where Events Include Disease Progression or Relapse, Second Malignancy, or Death
Description: Primary analysis will be based 1-sided log rank test comparison of EFS curves between the 2 randomized arms per intention-to-treat principle. Progression is defined as an ≥50% increase of in the product of the perpendicular diameters of any of the involved nodes or nodal masses or focal organ lesions in sites that were persistently PET positive; or recurrent PET positive lesions (Deauville 4, 5) in sites that had previously been PET negative regardless of change of size, as was the development of new PET avid measurable lesion(s) >1.5cm in any axis, or new sites of assessable disease. Relapse is defined in patients who achieved a prior CR but subsequently has an increase of ≥50% of the PPD in prior nodal or extranodal sites in a recurrently PET positive lesion(s), or the development of new measurable lesion(s) >1.5cm in any axis, or new sites of assessable disease. Second malignancy is defined based on report of a cancer that is not considered to be classic Hodgkin Lymphoma.
Time Frame: Up to 48 months after the last enrollment
Population: All the eligible patients who had undergone randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (ABVE-PC) | ARM II (Bv-AVEPC)
Number analyzed (Participants) | 289 | 298
percentage of participants | 82.5 [77.4 to 86.5] | 92.1 [88.4 to 94.7]
Statistical Analysis 1: Comparison: Arm I (ABVE-PC) vs ARM II (Bv-AVEPC); Assuming a 3-year EFS of 82% (5-year EFS of 78.4%, long term EFS of 76%) for standard arm, the study will have approximately 86% power for detecting an 8% improvement in 3-year EFS in the Bv-AVEPC arm (3-year EFS of 90%, 5-year EFS of 88.0%, long term EFS of 86.7%) in log rank test; Test type: Superiority; p = 0.0001, Log Rank; Used a one-sided log-rank test between 2 arms

2. Secondary Outcome: Percentages of Patients With Early Response Defined as no Slow Responding Lesions (SRL) and no Progressive Disease (PD) at Any Disease Sites Determined by Positron Emission Tomography (PET) Per Deauville Criteria Through Central Review
Description: The percentages of patients (with available PET scan) with no SRL and no PD will be compared between the two randomized arms to see if brentuximab vedotin in the chemotherapy backbone of doxorubicin hydrochloride, vincristine sulfate, etoposide, prednisone and cyclophosphamide (Bv-AVEPC) arm has a higher rate of early response compared to doxorubicin hydrochloride, bleomycin sulfate, vincristine sulfate, etoposide, prednisone, and cyclophosphamide (ABVE-PC) arm. Two-sample Z test of proportions at 1-sided alpha level of 0.05 will be used for these comparisons.
Time Frame: After 42 days of chemotherapy
Population: All the eligible patients who had undergone randomization and had PET result by central review after completed cycle 2
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm I (ABVE-PC) | ARM II (Bv-AVEPC)
Number analyzed (Participants) | 285 | 292
Percentage of patients | 80.7 [76.1 to 85.3] | 81.2 [76.7 to 85.7]

3. Secondary Outcome: Percentages of Patients Experiencing Grade 3+ Peripheral Neuropathy Assessed by Modified Balis Scale
Description: The percentages of patients experiencing grade 3+ peripheral neuropathy assessed by the treating clinician using the modified Balis scale. The "Modified Balis scale of Pediatric Neuropathy" allows clinicians to assign a score for sensory or motor neuropathy symptoms separately. Scores range from 1 to 4 with 1 being the least symptomatic state and 4 indicating a severe debility. The percentages of patients (with a score >/=3) will be compared between the 2 arms by two-sample Z test at 1-sided alpha level of 0.05.
Time Frame: From the enrollment of the patient to the time of analysis or the last follow-up; an average of 3.6 years.
Population: All the eligible patients who had undergone randomization
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm I (ABVE-PC) | ARM II (Bv-AVEPC)
Number analyzed (Participants) | 289 | 298
Percentage of patients | 5.5 [2.90 to 8.17] | 6.7 [3.87 to 9.55]

4. Other Pre Specified Outcome: Childhood International Prognostic Score (CHIPS) Score
Description: CHIPS will be computed for all patients and summarized by descriptive statistics. Will examine the association between CHIPS and early response by cross-tabulations and Chi-square tests within each arm separately, as well as logistic regression model where early response is the outcome variable and CHIPS the predictor variable combining the 2 arms with adjustment for randomized chemotherapy.
Time Frame: Baseline
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Dose of Radiation Received by Normal Tissues Following Chemotherapy on Either Study Arm
Description: Descriptive statistics will be used to summarize RT doses received by normal tissues on this study. Two-sample t-test will be used to compare the doses received on this study to those on prior studies.
Time Frame: Up to 48 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Efficacy of Involved Site Radiotherapy (ISRT) by Analyzing the Event-free Survival of Patients Treated With Response-adapted ISRT and by Evaluating Patterns of Relapse Following ISRT
Description: EFS for patients on each arm as well as those receiving ISRT or those with slow early response (SER) on each arm will be estimated. One-sample log rank test will be used to compare the observed EFS to the assumed baseline of 82% at 3 years to see if the observed EFS is significantly lower than the projection in these subsets.
Time Frame: Up to 3 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Risk of Relapse Among RRL Subjects That Have at Least One Lesion That is Deauville 3 at PET 2
Description: The risk of relapse for cases that are RRL, but have Deauville 3 lesions, will be compared to those that are classified as complete metabolic response at PET2 with solely Deauville 1 or 2 lesions with K-sample test.
Time Frame: Up to 48 months after the last enrollment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Pharmacokinetic (PK) Analyses
Description: PK concentration time profile will be evaluated.
Time Frame: Pre-dose and end of infusion on day 1, days 2, 3, 8, and 15 of cycle 4 and pre-dose on day 1 and day 22 of cycle 5 (each cycle = 21 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the enrollment of the patient to the time of analysis or the last follow-up; an average of 3.6 years. Ineligible patients are excluded. 5 patients (Arm I: 2 patients; Arm II: 3 patients) were also excluded from adverse events reporting due to never receiving any treatment, but their mortality status was observed. All-Cause Mortality includes all deaths collected on the study.
Description: Adverse Events are collected using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). Per the protocol, SAE reporting requirements and expedited reporting of AEs did differ for the Bv-AVEPC arm, given that Bv was under IND. All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table.
Arm/Group | Arm I (ABVE-PC) | ARM II (Bv-AVEPC)
All-Cause Mortality (participants affected / at risk) | 4/289 | 2/298
Serious Adverse Events (participants affected / at risk) | 11/287 | 66/295
Other Adverse Events (participants affected / at risk) | 206/287 | 209/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (ABVE-PC) (N=287) | ARM II (Bv-AVEPC) (N=295)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 9 (9)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 6 (6)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 6 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 2 (2)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1) | 3 (3)
Bone infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 6 (6)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 4 (4)
Platelet count decreased (Investigations) | 0 (0) | 2 (2)
Serum amylase increased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Muscle weakness left-sided (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 6 (6)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 4 (4) | 10 (10)
Thromboembolic event (Vascular disorders) | 0 (0) | 9 (9)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (ABVE-PC) (N=287) | ARM II (Bv-AVEPC) (N=295)
Anemia (Blood and lymphatic system disorders) | 89 (89) | 107 (107)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 90 (90) | 83 (83)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 2 (2)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 22 (22) | 28 (28)
Nausea (Gastrointestinal disorders) | 6 (6) | 10 (10)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Typhlitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 11 (11)
Fever (General disorders) | 6 (6) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 15 (15) | 7 (7)
Anaphylaxis (Immune system disorders) | 10 (10) | 7 (7)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2)
Arteritis infective (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 4 (4) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 4 (4)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 4 (4) | 7 (7)
Infective myositis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 3 (3)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 3 (3)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 7 (7) | 2 (2)
Shingles (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 4 (4) | 4 (4)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Vaginal infection (Infections and infestations) | 2 (2) | 0 (0)
Vulval infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 8 (8) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Alanine aminotransferase increased (Investigations) | 10 (10) | 11 (11)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (3)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (2)
Carbon monoxide diffusing capacity decreased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 2 (2)
GGT increased (Investigations) | 2 (2) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 3 (3)
Lymphocyte count decreased (Investigations) | 75 (75) | 71 (71)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 116 (116) | 144 (144)
Platelet count decreased (Investigations) | 81 (81) | 95 (95)
Serum amylase increased (Investigations) | 1 (1) | 1 (1)
Vital capacity abnormal (Investigations) | 2 (2) | 1 (1)
Weight gain (Investigations) | 1 (1) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 103 (103) | 121 (121)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 19 (19) | 13 (13)
Hyponatremia (Metabolism and nutrition disorders) | 9 (9) | 8 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 3 (3)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 28 (28) | 13 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 43 (43) | 42 (42)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 2 (2) | 1 (1)
Seizure (Nervous system disorders) | 3 (3) | 0 (0)
Syncope (Nervous system disorders) | 8 (8) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Premature menopause (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 11 (11) | 1 (1)
Thromboembolic event (Vascular disorders) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT02166463/Prot_SAP_000.pdf